CLINICAL TRIAL: NCT05748613
Title: Treatment of Stress and Anxiety in Mild Cognitive Impairment/Mild Alzheimer's Disease and Related Dementias - RCT
Brief Title: Anxiety Sensitivity Treatment to Reduce Anxiety in Alzheimer's
Acronym: ASTRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Ohio State University (Other); Ohio University (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Ph.D., Distinguished Research Professor, Department Chair, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00003432
Record Dates: First submitted 2023-02-07; First posted 2023-03-01 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Anxiety; Mild Cognitive Impairment; Alzheimer Disease; Dementia
Keywords: Computerized Intervention; Brief Treatment; Psychoeducation; Interoceptive Exposure; Older Adults; Care Partner; Anxiety Sensitivity
MeSH Terms: conditions — Anxiety Disorders; Cognitive Dysfunction; Alzheimer Disease; Dementia | interventions — NDC80 protein, human

STUDY DESIGN:
Intervention Model Description: Variable-sized permuted block randomization will be used to allocate participants to treatment condition, stratified by dementia severity (MCI vs. mild ADRD) and gender.
Who Masked: Participant, Outcomes Assessor
Masking Description: An independent assessor (blind to treatment condition) will conduct pre-intervention and follow-up assessments. The assessor will have extensive training and experience in conducting the relevant assessments including clinical interviews and neuropsychological evaluations. A separate interventionist will assist in the delivery of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Computerized Anxiety Sensitivity Treatment (Experimental): CAST is a transdiagnostic cognitive behavioral therapy (CBT)-based protocol designed to address elevated anxiety sensitivity (AS), particularly the amplification of cognitive stress symptoms including perceived confusion and memory problems. CAST is a fully computerized, 1-hour intervention containing video animation and audio narration throughout, as well as interactive features (e.g., brief quizzes to promote comprehension, introduction and practice with interoceptive exposures). Procedures draw heavily on standard CBT techniques; AS, a core vulnerability for anxiety and depression is targeted using these procedures. In CAST, participants are informed that "the primary purpose of the presentation is to highlight healthier, more productive, and effective ways of dealing with stress." Through participation in the intervention, people learn adaptive long-term strategies for tolerating, coping with, and effectively reducing distress and negative emotions.
  Interventions: Behavioral: Computerized Anxiety Sensitivity Treatment
- Health Education Control (Placebo Comparator): HEC is a fully computerized 1-hour control condition focused on increasing healthy behaviors and decreasing unhealthy behaviors. Content includes healthy eating, hydration, sleep and rest, exercise, stress management as well as other healthy lifestyle tips. To match the interactive components in the CAST condition, behavior tracking and goal-setting are included in HEC. The HEC protocol has been used in prior studies as a control condition for CAST to account for intervention modality and time. HEC is perceived positively, with high rates of acceptability. Importantly, HEC is inert with respect to the proposed mechanism of action (AS).
  Interventions: Behavioral: Health Education Control

INTERVENTIONS:
Behavioral: Computerized Anxiety Sensitivity Treatment — Brief computerized treatment for anxiety sensitivity
  Other Names: CAST
  Arms: Computerized Anxiety Sensitivity Treatment
Behavioral: Health Education Control — Brief computerized presentation on healthy behaviors
  Other Names: HEC, Physical Health Education Training ,PHET
  Arms: Health Education Control

SUMMARY:
The goal of this clinical trial is to test the effectiveness of a computerized anxiety sensitivity treatment (CAST) compared to a health education control (HEC) in older adults with mild cognitive impairment (MCI) or mild Alzheimer's Disease and related dementias (ADRD) and their care partners. The main questions it aims to answer are:

1. Efficacy of CAST in reducing anxiety and related symptoms among those with MCI/mild ADRD
2. Efficacy of CAST in reducing care partner burden among care partners of people living with MCI/mild ADRD
3. Explore treatment mechanisms using a multi-modal assessment battery of anxiety sensitivity and anxiety

Participants will complete six in-person visits including a baseline assessment, two intervention sessions, and three follow-up assessments at 1, 3, and 6-months posttreatment. Participants will also complete three weeks of ecological momentary assessments (EMAs) for one week prior to intervention, one week between intervention sessions, and one week after intervention.

If there is a comparison group: Researchers will compare CAST to HEC to see if CAST reduces anxiety and related symptoms in older adults with MCI/mild ADRD and care partner burden to a greater degree than HEC.

DETAILED DESCRIPTION:
Participants are dyads consisting of an older adult with MCI/mild ADRD and their care partner. Baseline assessment will include a neuropsychological evaluation to confirm cognitive status for the older adult with MCI/mild ADRD, a series of baseline questionnaires, and introduction to the EMA application. Dyads are randomized to either the CAST or HEC conditions. During CAST sessions, dyads view the CAST presentation and complete interoceptive exposures. An interventionist guides dyads through these sessions. During HEC, dyads view the HEC presentation and complete behavior tracking and goal-setting with the guidance of an interventionist. At both intervention sessions, dyads complete questionnaires including post assessments at the end of intervention session two. For the week prior to intervention session one, the week between the two intervention sessions, and the week after intervention session two, dyads complete daily EMAs about emotional and other factors using an application downloaded on a phone or tablet. At 1, 3, and 6-months follow-up assessments, dyads complete follow-up cognitive testing and outcome questionnaires.

ELIGIBILITY:
Inclusion Criteria:

DYAD

* Patient age 60+
* Care partner 18+
* Has care partner who will participate ("someone you have a reciprocal relationship with who provides you with emotional or physical support and helps with decision-making. This could be a spouse or significant other, relative, or close friend whom you spend a significant amount of time with.")
* Has smartphone or access to Wi-Fi

EITHER

* Score of 20 or above on the PROMIS-Anxiety short form (patient only) OR
* Score of 5 or above on SSASI (patient only) OR
* Score of 31 or above on NIH Toolbox Perceived Stress Scale score (patient only)

AND EITHER

1. Participant MoCA score is between 17 to 26

   OR
2. Participant Memory Complaint Scale score 3 or greater

   OR
3. Care partner quick dementia rating scale score between 2 to 12.5

Exclusion Criteria:

PATIENT

* Issues with seeing or hearing that would prevent reading or listening to computer presentations
* Medical conditions that would preclude participation in study
* Severe mental illness (e.g., schizophrenia, unmedicated bipolar disorder)

CARE PARTNER

* Issues with seeing or hearing that would prevent reading or listening to computer presentations
* Medical conditions that would preclude participation in study
* Severe mental illness (e.g., schizophrenia, unmedicated bipolar disorder)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety sensitivity pre intervention to posttreatment. | Baseline to immediately after the intervention
  Anxiety sensitivity will be measured using the Anxiety Sensitivity Index-3 (ASI-3). The ASI-3 is an 18-item self report measure with possible scores ranging from 0 to 72. Higher scores indicate higher anxiety sensitivity.
Change in anxiety pre intervention to 1-month follow-up. | Baseline to 1-month follow-up
  Anxiety will be assessed using the Patient-Reported Outcomes Measurement Information System - Anxiety (PROMIS Anxiety) Short Form 8a self-report measure. The PROMIS Anxiety is an 8-item self report questionnaire with possible scores ranging from 8 to 40. Higher scores indicate more anxiety.

SECONDARY OUTCOMES:
Change in negative affect pre intervention to 1-month follow-up. | Baseline to 1-month follow-up
  Negative affect will be assessed using the Positive and Negative Affect Schedule - Negative Affect (PANAS-NA). PANAS-NA is a 10-item self-report measure with possible scores ranging from 10 to 50. Higher scores indicate more negative affect.
Change in stress pre intervention to 1-month follow-up. | Baseline to 1-month follow-up
  Stress will be assessed with the NIH Toolbox - Perceived Stress. The NIH Toolbox - Perceived Stress is a 10-item self-report measure with possible scores ranging from 10 to 50. Higher scores indicate more stress.
Change in quality of life pre intervention to 1-month follow-up. | Baseline to 1-month follow-up
  Quality of life will be assessed with the NIH Toolbox General Life Satisfaction scale. The NIH Toolbox General Life Satisfaction scale is a 5-item self-report measure with possible scores ranging from 5 to 35. Higher scores indicate higher life satisfaction.
Change in depression pre intervention to 1-month follow-up. | Baseline to 1-month follow-up
  Depression will be assessed using the PROMIS - Depression Short Form 8b. The PROMIS - Depression is an 8-item self-report measure with possible scores ranging from 8 to 40. Higher scores indicate higher level of depression.
Change in cognitive functioning pre intervention to 1-month follow-up. | Baseline to 1-month follow-up
  Cognitive functioning will be assessed using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). RBANS assesses cognitive functioning in the following domains: immediate memory, visuospatial functioning, attention, language, and delayed memory.
Stability of anxiety sensitivity from posttreatment to 6-month follow-up. | Immediately after the intervention to 6-month follow-up.
  Anxiety sensitivity will be measured using the Anxiety Sensitivity Index-3 (ASI-3). The ASI-3 is an 18-item self report measure with possible scores ranging from 0 to 72. Higher scores indicate higher anxiety sensitivity.
Stability of anxiety from 1-month follow-up to 6-month follow-up. | 1-month to 6-month follow-up
  Anxiety will be assessed using the Patient-Reported Outcomes Measurement Information System - Anxiety (PROMIS Anxiety) Short Form 8a self-report measure. The PROMIS Anxiety is an 8-item self report questionnaire with possible scores ranging from 8 to 40. Higher scores indicate more anxiety.
Stability of depression from 1-month follow-up to 6-month follow-up. | 1-month to 6-month follow-up
  Depression will be assessed using the PROMIS - Depression Short Form 8b. The PROMIS - Depression is an 8-item self-report measure with possible scores ranging from 8 to 40. Higher scores indicate higher level of depression.
Stability of negative affect from 1-month follow-up to 6-month follow-up. | 1-month to 6-month follow-up
  Negative affect will be assessed using the Positive and Negative Affect Schedule - Negative Affect (PANAS-NA). PANAS-NA is a 10-item self-report measure with possible scores ranging from 10 to 50. Higher scores indicate more negative affect.
Stability of stress from 1-month follow-up to 6-month follow-up. | 1-month to 6-month follow-up
  Stress will be assessed with the NIH Toolbox - Perceived Stress. The NIH Toolbox - Perceived Stress is a 10-item self-report measure with possible scores ranging from 10 to 50. Higher scores indicate more stress.
Stability of quality of life from 1-month follow-up to 6-month follow-up. | 1-month to 6-month follow-up
  Quality of life will be assessed with the NIH Toolbox General Life Satisfaction scale. The NIH Toolbox General Life Satisfaction scale is a 5-item self-report measure with possible scores ranging from 5 to 35. Higher scores indicate higher life satisfaction.
Stability of cognitive functioning from 1-month follow-up to 6-month follow-up. | 1-month to 6-month follow-up
  Cognitive functioning will be assessed using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). RBANS assesses cognitive functioning in the following domains: immediate memory, visuospatial functioning, attention, language, and delayed memory.
Change in care partner burden from pre intervention to 1-month follow-up. | Baseline to 1-month follow-up
  Care partner burden will be assessed using the Zarit Burden Interview - Short. The Zarit Burden Interview - Short is a 12-item self-report questionnaire with a possible score range of 0 to 48. Higher scores indicate higher burden levels.
Change in objective measure of interoceptive fear conditioning pre to posttreatment | Baseline to immediately after the intervention
  Interoceptive fear conditioning will be assessed with a skin conductance response (SCR) during an interoceptive exposure. Higher SCR numbers indicate higher interoceptive fear.
Change in Loneliness from pre intervention to 1-month follow up | Baseline through Month 1 follow up
  Loneliness will be measured using the 10-item UCLA Loneliness Short form questionnaire. This self-report scale yields scores between 10 to 40 with higher scores indicating more significant loneliness symptoms.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Anxiety and Behavioral Health Clinic, Tallahassee, Florida
  - Ohio University, Athens, Ohio
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Zvolensky MJ, Garey L, Fergus TA, Gallagher MW, Viana AG, Shepherd JM, Mayorga NA, Kelley LP, Griggs JO, Schmidt NB. Refinement of anxiety sensitivity measurement: The Short Scale Anxiety Sensitivity Index (SSASI). Psychiatry Res. 2018 Nov;269:549-557. doi: 10.1016/j.psychres.2018.08.115. Epub 2018 Aug 29. PMID 30199696
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Vale FAC, Balieiro AP Jr, Silva-Filho JH. Memory complaint scale (MCS). Proposed tool for active systematic search. Dement Neuropsychol. 2012 Oct-Dec;6(4):212-218. doi: 10.1590/S1980-57642012DN06040004. PMID 29213800
- [Background] Galvin JE. THE QUICK DEMENTIA RATING SYSTEM (QDRS): A RAPID DEMENTIA STAGING TOOL. Alzheimers Dement (Amst). 2015 Jun 1;1(2):249-259. doi: 10.1016/j.dadm.2015.03.003. PMID 26140284
- [Background] Randolph C, Tierney MC, Mohr E, Chase TN. The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): preliminary clinical validity. J Clin Exp Neuropsychol. 1998 Jun;20(3):310-9. doi: 10.1076/jcen.20.3.310.823. PMID 9845158
- [Background] Delis, D. C., Kaplan, E., & Kramer, J. H. (2001). Delis-Kaplan Executive Function System (D-KEFS) [Database record]. APA PsycTests.
- [Background] Wechsler, D. (2008). Wechsler Adult Intelligence Scale--Fourth Edition (WAIS-IV) [Database record]. APA PsycTests.
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Taylor S, Zvolensky MJ, Cox BJ, Deacon B, Heimberg RG, Ledley DR, Abramowitz JS, Holaway RM, Sandin B, Stewart SH, Coles M, Eng W, Daly ES, Arrindell WA, Bouvard M, Cardenas SJ. Robust dimensions of anxiety sensitivity: development and initial validation of the Anxiety Sensitivity Index-3. Psychol Assess. 2007 Jun;19(2):176-88. doi: 10.1037/1040-3590.19.2.176. PMID 17563199
- [Background] Kupst MJ, Butt Z, Stoney CM, Griffith JW, Salsman JM, Folkman S, Cella D. Assessment of stress and self-efficacy for the NIH Toolbox for Neurological and Behavioral Function. Anxiety Stress Coping. 2015;28(5):531-44. doi: 10.1080/10615806.2014.994204. Epub 2015 Feb 10. PMID 25577948
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Craig, C., Marshall, A., Sjostrom, M., Bauman, A., Lee, P., Macfarlane, D., ... & Stewart, S. (2017). International physical activity questionnaire-short form. J Am Coll Health, 65(7), 492-501.
- [Background] Zarit, S., Orr, N. K., & Zarit, J. M. (1985). The hidden victims of Alzheimer's disease: Families under stress. NYU press.
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Hughes CP, Berg L, Danziger WL, Coben LA, Martin RL. A new clinical scale for the staging of dementia. Br J Psychiatry. 1982 Jun;140:566-72. doi: 10.1192/bjp.140.6.566. PMID 7104545
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Hatcher, R. L., & Gillaspy, A. (2006). Working Alliance Inventory-Short Revised [Database record]. APA PsycTests.
- [Derived] Markley AE, Stratton KM, Cho GY, Schmidt NB, Suhr J, Sheffler JL, Nguyen C, Schubert FT, Quiles JRG, Potter MR, Meynadasy MA, Irvin SM, Allan NP. Study design and protocol for cognitive anxiety sensitivity treatment for anxiety in adults with mild cognitive impairment or dementia. Contemp Clin Trials. 2025 Sep;156:108044. doi: 10.1016/j.cct.2025.108044. Epub 2025 Aug 6. PMID 40774425